CLINICAL TRIAL: NCT04221555
Title: Neoadjuvant Durvalumab (MEDI4736) Plus Docetaxel, Oxaliplatin, S-1 (DOS) Followed by Surgery and Adjuvant Durvalumab Plus S-1 Chemotherapy in Potentially Resectable MMR Proficient (pMMR) Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma
Brief Title: Trial of Neoadjuvant Durvalumab Plus Docetaxel, Oxaliplatin, S-1 Followed by Surgery and Adjuvant Durvalumab Plus S-1 Chemotherapy in Potentially Resectable MMR Proficient Gastric or Gastroesophageal Junction Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Min-Hee Ryu, Professor, Asan Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC2001
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Resectable Gastric or Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — Docetaxel; Oxaliplatin; S 1 (combination); durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- the main treatment group (Experimental): pMMR tumor
  Interventions: Drug: Docetaxel, Oxaliplatin, S-1 and Durvalumab
- the exploratory group (Active Comparator): dMMR tumor
  Interventions: Drug: Durvalumab and Tremelimumab

INTERVENTIONS:
Drug: Docetaxel, Oxaliplatin, S-1 and Durvalumab — 1. Neoadjuvant treatment Durvalumab 1120 mg IV on day (D) 1, Docetaxel 50 mg/m2 intravenously (IV) on D1, oxaliplatin 100 mg/m2 IV on D1, S-1 40 mg/m2 bid orally on D1-14, will be administered every three weeks for three cycles.
  2. Surgery
  3. Adjuvant treatment After 4-6 weeks from surgery, S-1 40 mg/m2 bid orally on D1-28 plus durvalumab 1120 mg on D1 and D22 will be administered every 6 weeks for 12 months as an adjuvant treatment.
  Arms: the main treatment group
Drug: Durvalumab and Tremelimumab — 1. Neoadjuvant treatment Durvalumab 1500 mg IV and tremelimumab 75 mg IV on D1 will be administered every four weeks for three cycles.
  2. Surgery
  3. Adjuvant treatment After 4-6 weeks from surgery, durvalumab 1500 mg on D1 will be administered every 4 weeks for 12 months as an adjuvant treatment.
  Arms: the exploratory group

SUMMARY:
Neoadjuvant durvalumab (MEDI4736) plus docetaxel, oxaliplatin, S-1 (DOS) followed by surgery and adjuvant durvalumab plus S-1 chemotherapy in potentially resectable MMR proficient (pMMR) gastric or gastroesophageal junction (GEJ) adenocarcinoma

DETAILED DESCRIPTION:
* Treatment for the main treatment group (pMMR tumor)

  1. Neoadjuvant treatment Durvalumab 1120 mg IV on day (D) 1, Docetaxel 50 mg/m2 intravenously (IV) on D1, oxaliplatin 100 mg/m2 IV on D1, S-1 40 mg/m2 bid orally on D1-14, will be administered every three weeks for three cycles.
  2. Surgery
  3. Adjuvant treatment After 4-6 weeks from surgery, S-1 40 mg/m2 bid orally on D1-28 plus durvalumab 1120 mg on D1 and D22 will be administered every 6 weeks for 12 months as an adjuvant treatment.
* Treatment for the exploratory group (dMMR tumor)

  1. Neoadjuvant treatment Durvalumab 1500 mg IV and tremelimumab 75 mg IV on D1 will be administered every four weeks for three cycles.
  2. Surgery
  3. Adjuvant treatment After 4-6 weeks from surgery, durvalumab 1500 mg on D1 will be administered every 4 weeks for 12 months as an adjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed pathologically proven potentially resectable gastric or GEJ adenocarcinoma
2. Clinical stages of T3-4N0 or T2-4N+ according to the American Joint Committee on Cancer (AJCC) 8th edition by computed tomography (CT)
3. Microsatellite-instability (MSI) status determined by immunohistochemical (IHC) staining
4. No peritoneal seeding identified by laparoscopy if suspected by CT
5. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations
6. Age > 18 years at time of study entry
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
8. Life expectancy of > 12 months
9. Body weight > 30kg
10. No existing neuropathy
11. Adequate normal organ and marrow function as defined below:

    * Haemoglobin ≥9.0 g/dL
    * Absolute neutrophil count (ANC) 1.5 (or 1.0) x (> 1500 per mm3)
    * Platelet count ≥100 (or 75) x 109/L (>75,000 per mm3)
    * Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN)
    * AST (SGOT)/ALT (SGPT) ≤2.5 x institutional ULN
    * Measured creatinine clearance (CL) > 40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:
12. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause.
13. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up

Exclusion Criteria:

1. Participation in another clinical study with an investigational product during the last 2 weeks
2. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
3. Any concurrent chemotherapy, immunotherapy, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacementtherapy) is acceptable
4. Major surgical procedure within 28 days prior to the first dose of durvalumab
5. Distant metastasis including M1 lymph node
6. Unable to take medication orally
7. Gastric outlet obstruction and/or severe gastrointestinal bleeding
8. Impaired bowel absorption, including any of the following:

   * Bowel obstruction
   * Chronic inflammatory bowel disease
   * History of extended bowel resection
   * Gastric dumping syndrome
9. History of allogenic organ transplantation
10. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    * Patients with vitiligo or alopecia
    * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
    * Any chronic skin condition that does not require systemic therapy
    * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
    * Patients with celiac disease controlled by diet alone
11. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events (AEs) or compromise the ability of the patient to give written informed consent
12. History of another primary malignancy except for

    * Malignancy treated with curative intent and with no known active disease ≥ 5 years before the first dose of durvalumab and of low potential risk for recurrence
    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    * Adequately treated carcinoma in situ without evidence of disease
13. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart)
14. History of active primary immunodeficiency
15. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
16. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
    * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
17. Receipt of live attenuated vaccine within 30 days prior to the first dose of durvalumab. Note: Patients, if enrolled, should not receive live vaccine whilst receiving durvalumab and up to 30 days after the last dose of durvalumab
18. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab
19. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients
20. Prior randomisation or treatment in a previous durvalumab or tremelimumab clinical study regardless of treatment arm assignment

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2020-05-13 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete regression (pCR) rate | 3 years

SECONDARY OUTCOMES:
R0 resection rate | 3 years
Disease free survival (DFS) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Min-Hee Ryu, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea